CLINICAL TRIAL: NCT05936138
Title: A Phase 1, Parallel, Single-Dose, Open-Label, Single-Period Study of LY3502970 in Participants With Normal Renal Function and Participants With Renal Impairment
Brief Title: A Study of LY3502970 in Participants With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18633; J2A-MC-GZPC (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3502970 (Control) (Experimental): LY3502970 administered orally to participants with normal renal function
  Interventions: Drug: LY3502970
- LY3502970 (Severe Renal Impairment) (Experimental): LY3502970 administered orally to participants with severe renal impairment
  Interventions: Drug: LY3502970
- LY3502970 (End-Stage Renal Disease) (Experimental): LY3502970 administered orally to participants with end-stage renal disease (ESRD)
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to assess the amount of study drug (LY3502970) that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment compared to participants with normal renal function. The safety and tolerability of LY3502970 will also be evaluated in these participants. The study will last up to 6 weeks including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index within the range 18.5 to 42.0 kilograms per meter squared (kg/m²), inclusive.
* Men and women who agree to use highly effective or effective methods of contraception may participate in this trial.

Participants with Normal Renal Function:

* Healthy males or females as determined by medical history, physical examination, and other screening procedures, with normal renal function. Have estimated glomerular filtration rate (eGFR) of greater than or equal to 90 milliliter per minute (mL/min)

Participants with Renal Impairment:

* Severe renal impairment: Have eGFR of 15 to 29 mL/min and not requiring hemodialysis.
* ESRD: Participants who have been on a stable hemodialysis schedule for at least 3 months prior to planned dosing.

Exclusion Criteria:

* Have a current, functioning organ transplant. Non-functional renal allografts may be allowed.
* Regularly use known drugs of abuse or show positive findings on urinary drug screen that are not otherwise explained by permitted concomitant medications.
* Have known allergies to LY3502970, related compounds, or any components of the formulation, or history of severe atopy.
* Are lactating, pregnant, or intend to become pregnant, or to breastfeed during the study.
* Have a history or presence of chronic or acute pancreatitis

Participants with Renal Impairment:

* Have hemoglobin <8.5 g/dL.
* Participants with Type 2 Diabetes Mellitus if they have taken any Glucagon-like Peptide-1 Receptor Agonists (GLP1-RA) or a Dipeptidyl Peptidase 4 (DPP4) inhibitor in the past 6 weeks or 5 half-lives prior to dosing, whichever is longer, prior to dosing on Day 1

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3502970 | Predose up to 12 days postdose
  PK: (AUC0-∞) of LY3502970
PK: Area under the concentration versus time curve from time zero to last time point (AUC0-tlast) of LY3502970 | Predose up to 12 days postdose
  PK: AUC0-tlast of LY3502970
PK: Maximum observed concentration (Cmax) of LY3502970 | Predose up to 12 days postdose
  PK: Cmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance For multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No